CLINICAL TRIAL: NCT04462237
Title: The Effect of Recombinant Human Platelet-derived Growth Factor in Combination With Collagen Matrix for the Treatment of Multiple Adjacent Gingival Recessions: A Randomized Clinical Trial
Brief Title: Recombinant Human Platelet-derived Growth Factor in Combination With Collagen Matrix
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Lorenzo Tavelli, Principal Investigator, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HUM00177214
Record Dates: First submitted 2020-06-29; First posted 2020-07-08 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Gingival Recession; Platelet Derived Growth Factor
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- collagen matrix + platelet-derived growth factor (Experimental): Root coverage procedure using collagen matrix + platelet-derived growth factor for the treatment of multiple adjacent gingival recessions
  Interventions: Procedure: Root coverage procedures
- collagen matrix alone (Active Comparator): Root coverage procedure using collagen matrix alone (without the use of the platelet-derived growth factor) for the treatment of multiple adjacent gingival recessions
  Interventions: Procedure: Root coverage procedures

INTERVENTIONS:
Procedure: Root coverage procedures — Treatment of multiple adjacent gingival recession using a coronally advanced flap

SUMMARY:
The present randomized clinical trial is aimed at evaluating the efficacy of recombinant human platelet-derived growth factor in combination with collagen matrix for the treatment of multiple adjacent gingival recessions

DETAILED DESCRIPTION:
Despite the fact that gingival recession is most often a generalized condition rather than being localized to a single tooth, most of the data currently found in the literature pertains to the treatment of localized gingival recessions.

The gold standard treatment for this condition involves the use of an autogenous connective tissue graft, that is associated with increased patient morbidity.

Biomaterials have progressively gained popularity due to their advantages when compared to autogenous grafts, such as unrestricted availability, avoidance of a secondary surgical site, reduction of the surgical time, and the patient's preference.

Collagen matrix is one of the most used soft tissue substitute for the treatment of gingival recessions. Combining this scaffold material with a growth factor could enhance its outcomes. In particular, root coverage using platelet-derived growth factor can also promote regeneration of new cementum, periodontal ligament and bone.

Therefore, the aim of the present study is to investigate the effect of platelet-derived growth factor in combination with collagen matrix outcomes for the treatment of multiple adjacent gingival recessions.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Periodontally and systemically healthy
* Full-mouth plaque score and full-mouth bleeding score ≤ 20% (measured at four sites per tooth)
* At least two multiple adjacent gingival recessions (with at least one 2 mm or deeper) requiring surgical intervention for root coverage
* No interproximal attachment/bone loss
* No prior experience of root coverage procedures within the last 1 year
* The patient must be able to perform good oral hygiene

Exclusion Criteria:

* Contraindications for periodontal surgery
* Patients pregnant or attempting to get pregnant (self-reported)
* Untreated periodontitis
* Persistence of uncorrected gingival trauma from traumatic toothbrushing
* Interdental attachment loss greater than 1 mm or furcation involvement in the teeth to be treated
* Presence of severe tooth malposition, rotation or clinically significant super-eruption
* Self-reported current smoking more than 10 cigarettes/day or pipe or cigar smoking
* Allergy to collagen-based medical products

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-09-09 (Actual); Primary Completion 2021-08-18 (Actual); Study Completion 2021-08-18 (Actual)

PRIMARY OUTCOMES:
Mean Root Coverage | 6 months
  amount of recession reduction compared to the baseline recession depth
Keratinized tissue width gain | 6 months
  amount of keratinized tissue width gain from the baseline
Gingival thickness gain | 6 months
  amount of gingival thickness gain from the baseline

SECONDARY OUTCOMES:
3D volumetric changes | 6 months
  Soft tissue volumetric variation evaluated with digital softwares
Tissue perfusion variations | 6 months
  Tissue perfusion variations compared to baseline at the different follow-up using ultrasonography
Patient-related outcomes | 6 months
  Patient self reported perception of the procedure in terms of morbidity, satisfaction and esthetic outcomes. Visual analogue scales (from 0 to 100) will be used to assess these outcomes
Esthetic outcomes | 6 months
  evaluated using the root coverage esthetic score (from 0 to 10)

OTHER OUTCOMES:
Differences in Angiogenic Biomarkers | 3 months
  Within-subject difference between the concentrations at the control and test sites

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Tavelli, DDS, MS, Principal Investigator — University of Michigan; William Giannobile, DDS, MS, DMSc, Study Chair — University of Michigan; Hom-Lay Wang, DDS, MS, PhD, Study Director — University of Michigan
Locations (1):
- University of Michigan School of Dentistry, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tavelli L, Nguyen T, Rodriguez MV, Mancini L, Giannobile WV, Barootchi S. Tissue Perfusion and Biomarkers Assessment Following Root Coverage Procedures. J Periodontal Res. 2025 Nov;60(11):1117-1131. doi: 10.1111/jre.13374. Epub 2025 Jan 22. PMID 39843351
- [Derived] Tavelli L, Barootchi S, Rodriguez MV, Mancini L, Majzoub J, Travan S, Sugai J, Chan HL, Kripfgans O, Wang HL, Giannobile WV. Recombinant human platelet-derived growth factor improves root coverage of a collagen matrix for multiple adjacent gingival recessions: A triple-blinded, randomized, placebo-controlled trial. J Clin Periodontol. 2022 Nov;49(11):1169-1184. doi: 10.1111/jcpe.13706. Epub 2022 Jul 31. PMID 35871600